CLINICAL TRIAL: NCT03643510
Title: Phase II Study of Fulvestrant in Combination With Abemaciclib in Hormone Receptor Positive Adenocarcinoma of Endometrium
Brief Title: Evaluating Cancer Response to Treatment With Abemaciclib and Fulvestrant in Women With Recurrent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-107
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Adenocarcinoma of Endometrium
Keywords: Hormone Receptor Positive; Fulvestrant; Abemaciclib; 18-107
MeSH Terms: interventions — Fulvestrant; abemaciclib

STUDY DESIGN:
Intervention Model Description: This is a prospective, single arm study of combination CDK4 and CDK6 dual inhibitor Abemaciclib and selective estrogen receptor degrader Fulvestrant in hormone receptor positive recurrent endometrial carcinomas.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fulvestrant in Combination with Abemaciclib (Experimental): Eligible patients will take Abemaciclib 150 milligrams mg orally once every 12 hours on days 1-28. Fulvestrant will be dosed 500mg intramuscularly (IM) on days 1 and 15 during cycle 1 and then on Day 1 during subsequent cycles. Each cycle will be 28 days in duration. Patients will receive study treatment until disease progression, intolerable toxicity, elective withdrawal from the study, or study termination.
  Interventions: Drug: Fulvestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant will be dosed 500mg intramuscularly (IM) on days 1 and 15 during cycle 1 and then on Day 1 during subsequent cycles.
Drug: Abemaciclib — Abemaciclib 150 milligrams mg orally once every 12 hours on days 1-28.

SUMMARY:
The purpose of this study is to determine the effectiveness of the combination of abemaciclib and fulvestrant in treating this type of cancer and to determine the types and severity of side effects caused by treatment with abemaciclib and fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed an approved informed consent and authorization permitting release of personal information.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 AND Karnofsky Performance Status (KPS) ≥ 80
* Patients are not required to but may have received no more than two prior chemotherapeutic regimens for management of endometrial carcinoma (including adjuvant chemotherapy). Initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy.

  * Chemotherapy administered in conjunction with primary radiation as a radiosensitizer WILL be counted as a systemic chemotherapy regimen.
* Patients are not required to but may have received a single line of prior hormonal therapy with either an antiestrogen, anti-progesterone (or combination) or an aromatase inhibitor. Patients may not have received more than 1 line of endocrine therapy. This will not count toward prior therapy total.
* Resolution of adverse effects of recent surgery, radiotherapy, chemotherapy, or hormonal therapy to Grade ≤1 prior to first study treatment with the exception of peripheral neuropathy and alopecia.
* Postmenopausal status due to either surgical or natural menopause. Post-menopausal status due to surgical/natural menopause requires at least 1 of the following:

  * History of hysterectomy
  * Prior bilateral oophorectomy
  * Age ≥ 60
  * Age ≤ 60 and amenorrheic for at least 12 months (in the absence of chemotherapy, hormonal therapy or ovarian suppression) and FSH and estradiol levels in the postmenopausal range.
  * Have a negative serum pregnancy test at baseline (within 7 days prior to -initiation of treatment) and agree to use medically approved precautions to prevent pregnancy during the study and for 1 month following the last dose of Abemaciclib.
* For patients of childbearing potential, agreement to use two effective forms of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for the duration of the study and for 30 days after the last abemaciclib dose.
* Patients must agree to pre- and post-treatment tumor biopsies
* Disease that is measurable as per RECIST v1.1.

  * Tumors within a previously irradiated field wi ll be designated as "nontarget" lesions unless progression is documented, or a biopsy is obtained to confirm persistence of tumor ≥ 90 days following completion of radiation therapy.
* No active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection). Any hormonal therapy directed at the malignant tumor must be discontinued at least 2 weeks prior to the first study treatment.
* Patients must meet all the following criteria to be eligible for study entry:

  1. Patients must have recurrent or persistent endometrial carcinoma that is refractory to curative therapy or established treatments.
  2. Histologic confirmation of the original primary tumor is required.
  3. Histologic or cytologic confirmation of the recurrent/progressive disease is desired, but not required.
  4. Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, de-differentiated, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma.

     * For mixed epithelial cell type endometrial carcinomas, the endometrioid component should comprise at least 95% of the total tumor and the non-endometrioid component should comprise less than 5% of the total tumor.
  5. Patient must have hormone receptor positive (HR+) endometrial cancer confirmed by MSK pathology:

     * To fulfill the requirement for HR+ disease, tumor must express by immunohistochemistry (IHC), at least 1 of the hormone receptors (estrogen receptor [ER] or progesterone receptor [PgR] as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines (Hammond et al, 2010)
* Any prior therapy directed at the malignant tumor, including immunologic agents and radiotherapy, must be discontinued prior to first study treatment.

  * Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy).
  * Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 7 days prior to first study treatment:

  * Absolute neutrophil count (ANC) ≥1500/109dL
  * Platelet count ≥ 100,000/109dL
  * Hemoglobin ≥ 9.0 g/dL
  * Albumin ≥ 3.0 g/dL
  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
  * AST and ALT ≤ 3.0x ULN
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 xULN. For patients requiring therapeutic anticoagulation, a stable INR ≤3 x ULN is required.
* Are able to swallow capsules/tablets
* Are willing to follow study procedures
* For patients of childbearing potential, agreement to use two effective forms of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for the duration of the study and for 30 days after the last abemaciclib dose.

Exclusion Criteria:

* Patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization, or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study
* Patient who is experiencing a visceral crisis, lymphangitic disease spread, leptomeningeal carcinomatosis. Visceral crisis is not the mere presence of visceral metastases but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of disease.
* Patients who have received prior treatment with fulvestrant, everolimus, temsirolimus, ridaforolimus or another mTor inhibitor, or any CDK4 and CDK6 inhibitor.
* Patients who have received an autologous or allogenic stem-cell transplant.
* Clinically significant history of liver disease, including cirrhosis and current alcohol abuse.
* Patients who have active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection
* Presence of positive test results for hepatitis B (hepatitis B surface antigen [HBsAGg] and/or total HB core antibody [anti-HBc]) or hepatitis C (hepatitis C virus [HCV] antibody serology testing)
* Patients positive for anti-HBc are eligible only if also positive for HB surface antibody (anti-HBs) and polymerase chain reaction (PCR) assay is negative for HBV DNA.

  * Patients positive for HCV antibody are eligible only if testing for HCV RNA is negative.
* Known HIV infection.
* Active autoimmune disease that is not controlled by nonsteroidal anti -inflammatory drugs.
* Pregnancy, lactation, breastfeeding.
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure within 14 days prior to randomization, or significant traumatic injury within 28 days prior to Day 1 or anticipation of the need for major surgery during the course of study treatment.
* Have initiated biphosphonate or RANK ligand targeted agents (for example,denosumab) <7 days prior to Cycle 1 Day 1
* Uncontrolled hypomagnesemia or hypokalemia, defined as values below the lower limit of normal despite optimal electrolyte supplementation or management
* Leptomeningeal disease as a manifestation of cancer
* Known untreated or active central nervous system (CNS) metastases (progression or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteria:

  1. Presence of measurable disease outside the CNS
  2. No radiographic evidence of worsening upon the completion of CNSdirected therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
  3. No history of intracranial hemorrhage or spinal cord hemorrhage
  4. No ongoing requirement for dexamethasone as therapy for CNS disease (anticonvulsants at a stable dose are allowed)
  5. Screening CNS radiographic study is ≤ 6 months after most recent intervention for CNS metastases (neurological resection, radiotherapy, or brain biopsy) and ≥ 4 months after the discontinuation of corticosteroids
* Inability to comply with study and follow-up procedures
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the i nvestigator"s opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Patients who have:

  * History of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to ventricular tachycardia and ventricular fibrillation) or sudden cardiac arrest
  * New York Heart Association Class II or greater congestive heart failure (see Appendix A)
  * History of malabsorption syndrome or other condition that would interfere with enteral absorption
  * Inability or unwillingness to swallow pills
  * Serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial Cancer
Enrollment: 28 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 year
  defined as the percentage of patients with complete response (CR) + partial response (PR)]after initiating therapy. Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Green, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm